CLINICAL TRIAL: NCT07061275
Title: Telehealth-Supervised Resistance Training to Improve Functional Capacity and Muscle Strength in Children With Cerebral Palsy: Protocol for a Single-Arm Intervention Study
Brief Title: Telehealth-Supervised Resistance Training for Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Collaborators: Shanghai University of Sport (Other)
Responsible Party: Principal Investigator, Yang Zhang, Principle scientist, Hunan Normal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HunanNU-2025-506
Record Dates: First submitted 2025-06-25; First posted 2025-07-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: balance; cost; exercise training; gait; group exercise; rehabilitation; strength training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-arm interventional trial to evaluate the feasibility and efficacy of telehealth-supervised resistance training in children with mild CP. From an ethical standpoint, the use of a single-arm design is justified by the well-established benefits of resistance training for improving muscle morphology in this population. Prior RCT have also consistently shown that resistance training produces moderate to large improvements in functional capacity and mobility. Given this body of evidence, withholding treatment or assigning children to a non-intervention control group may present ethical concerns, particularly when a safe, home-based alternative is possibly available. Therefore, a single-arm design is both ethically sound and methodologically appropriate for addressing the research question.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth-Supervised Resistance Training (Experimental): The intervention consists of a 12-week telehealth-supervised resistance training program designed for children with mild CP. Training sessions will be conducted live via a secure smartphone-based streaming platform three times per week, with each session lasting approximately 40 minutes. Each session includes a 5-minute warm-up, 30 minutes of structured exercises, and a 5-minute cool-down period. Sessions are scheduled in the evening hours (around 7:00-8:00 PM) to accommodate children's school schedules and ensure caregiver availability during home-based participation.
  Interventions: Behavioral: Telehealth-Supervised Resistance Training

INTERVENTIONS:
Behavioral: Telehealth-Supervised Resistance Training — The exercise protocol will incorporate a variety of exercise modalities adapted for home use in limited space environments. Elastic resistance bands will be used for lower-limb strength exercises such as leg presses, hip abduction, and ankle dorsiflexion, while sandbag-style leg weights will be employed for activities including knee extensions, seated marches, and standing squats. To target balance, low-cost tools such as foam pads, balance cushions, or step platforms will be used for tasks including static standing, single-leg stance, and step-up exercises designed to challenge postural control in a safe, progressive manner.
  Sessions will be delivered through a secure live-streaming platform accessible on smartphones. The streaming platform supports background audio, allowing exercise sessions to be accompanied by music, which may help increase motivation and enjoyment for participating children. Each session will be led by trained instructors from the Hunan Normal University.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and potential benefits of telehealth-supervised resistance training in ambulatory children aged 6 to 15 years with cerebral palsy (CP) classified as Gross Motor Function Classification System (GMFCS) levels I-III.

The main questions it aims to answer are:

* Is a 12-week telehealth-delivered resistance training program feasible and acceptable for children with CP and their caregivers?
* Can the program improve physical function and psychosocial well-being in this population?

Participants will:

* Take part in three 40-minute, live-streamed resistance training sessions each week for 12 weeks, using elastic bands, sandbag weights, and balance tools
* Complete physical assessments before and after the program, including the 1-minute walk test, 10-meter walk test, 30-second sit-to-stand test, and Pediatric Balance Scale
* Complete quality of life surveys using the Pediatric Quality of Life Inventory (PedsQL™ 3.0 CP Module)
* Have caregivers complete a custom questionnaire about the cost and acceptability of the program

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a lifelong neurodevelopmental disorder caused by non-progressive disturbances in the developing fetal or infant brain. It is characterized by impairments in movement and posture, often accompanied by disturbances in sensation, perception, cognition, communication, and behavior. Globally, CP affects an estimated 17 million individuals, with a birth prevalence of approximately 2 to 2.5 per 1,000 live births . In China, more than 6 million children are estimated to be living with CP, and approximately 40,000 new cases occur each year.

Motor impairments in CP often lead to compromised gross motor function, altered gait mechanics, and reduced muscle force generation. These deficits significantly impact daily living activities, including walking, stair climbing, and performing transitions such as standing from a seated position. Muscle weakness, in particular, is a primary contributor to poor mobility and reduced participation in community and educational settings. Children with Gross Motor Function Classification System (GMFCS) levels I-III are ambulatory but may still experience fatigue, slow gait speed, or difficulty in navigating uneven terrain. Resistance training has gained empirical support as an effective intervention for improving muscle strength, joint stability, and gross motor function in children with mild CP. As highlighted in our recent meta-analysis, a growing body of evidence from randomized controlled trials indicates that well-structured, progressive resistance training programs lead to measurable improvements in lower-limb muscle morphology, which is directly related to strength, walking performance, and motor control. Ultimately, these muscle adaptations are closely linked to gains in functional independence, including stair climbing, transitions, and longer walking endurance - activities essential for participation in home, school, and recreational settings.

Despite its proven efficacy, access to therapist-supervised or facility-based resistance training remains limited for many families - particularly those living in low-resource or rural settings. Children with CP are disproportionately represented among lower-income households, and socioeconomic factors can severely limit access to regular rehabilitation services. Out-of-pocket expenses for transportation, time off work for caregivers, and session fees create significant burdens, contributing to inadequate adherence and suboptimal rehabilitation outcomes.

Telehealth has emerged as a promising strategy to overcome these barriers by delivering structured, therapist-guided interventions remotely. The expansion of digital health technologies, particularly during the COVID-19 pandemic, has accelerated the adoption of tele-rehabilitation for various clinical populations. Live-streamed and app-based exercise training programs have shown promise in able-bodied populations due to their low cost, flexibility, and minimal infrastructure requirements. For children with CP, a telehealth model may increase access and engagement while reducing logistical and financial strain on families.

To our knowledge, no published studies have systematically evaluated the effects of telehealth-supervised resistance training specifically targeting improvements in functional capacity among children with CP. Given the affordability of this model - tele-exercise classes may cost as little as 10 CNY per session, and home exercise kits can be assembled using low-cost elastic bands and resistance tools - this approach may provide a viable, family-centered solution. The model is particularly attractive in the context of China and other low- and middle-income countries, where rehabilitation access is highly variable and often concentrated in urban centers.

The present study aims to evaluate the feasibility and efficacy of a telehealth-supervised resistance training program targeting lower-limb muscle strength and functional capacity in children with mild CP. This single-arm intervention trial will examine changes in gross motor ability, lower-limb muscle function, and parent-reported outcomes following a 3-month remotely supervised exercise protocol. The findings will provide initial evidence to inform the scalability and cost-effectiveness of telehealth-based rehabilitation models and may offer an inclusive and sustainable approach for pediatric rehabilitation in socioeconomically disadvantaged settings.

ELIGIBILITY:
Inclusion Criteria:

* No history of heart disease or family history of heart disease;
* Children classified as GMFCS levels I, II, or III;
* Dependent on assistive mobility devices, such as wheelchairs or posture support walkers, for activities of daily living;
* Medically stable and able to sit upright for at least 30 minutes;
* Able to understand simple verbal or visual instructions.

Exclusion Criteria:

* Aged under 6 years or over 15 years;
* Received botulinum toxin A injections for lower limb muscles within six months prior to baseline assessment;
* Implanted with an intrathecal baclofen pump, or has a history of lower limb-related orthopedic or neurosurgical interventions (such as tendon lengthening, osteotomy, or selective dorsal rhizotomy);
* Has uncontrolled epilepsy, severe cognitive impairment, or other comorbidities.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
1-minute walk test | Baseline (week 0) and post-intervention (week 12)
  Participants will be instructed to walk as far as possible without running within one minute, and the total distance covered will be recorded.
10-meter walk test | Baseline (week 0) and post-intervention (week 12)
  Participants will be asked to walk as fast as possible for 10 meters. The test will be performed under two conditions - self-selected and fast walking speeds - with the average of three trials recorded per condition.
Lower-limb muscle strength | Baseline (week 0) and post-intervention (week 12)
  Lower-limb muscle strength will be assessed using the 30-second sit-to-stand test (30s STS), a simple, reliable functional test in which children are instructed to complete as many full STS repetitions as possible from a standard chair within 30 seconds (Romin et al., 2024).
Balance | Baseline (week 0) and post-intervention (week 12)
  Balance will be measured using the Pediatric Balance Scale, a 14-item assessment adapted from the Berg Balance Scale that evaluates functional postural control and is validated for ambulatory children with CP (Her et al., 2012). Tasks include standing on one foot, turning in place, and reaching forward
Pediatric Quality of Life Inventory | Baseline (week 0) and post-intervention (week 12)
  To assess life satisfaction and psychosocial well-being, children and their caregivers will complete the Pediatric Quality of Life Inventory™ (PedsQL) - Cerebral Palsy Module (Varni et al., 2006). This validated instrument measures multiple domains, including physical functioning, emotional well-being, and social participation. Both self-report and parent-proxy formats will be utilized for children aged 5-18 years.

SECONDARY OUTCOMES:
cost-acceptability survey | Post-intervention (week 12)
  Caregivers will complete a cost-acceptability survey designed to assess the perceived affordability and feasibility of the telehealth-delivered training model. The survey will include statements such as "The program is affordable for my family," "10 CNY per session is a fair price for the quality of the program," and "I would continue the training even if not reimbursed," rated on a 5-point Likert scale from strongly agree to strongly disagree. Caregivers will also answer an open-ended question: "What is the maximum price you would be willing to pay per session?" These items aim to evaluate the scalability and economic sustainability of this intervention from the perspective of end users.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhou, PhD, Study Director — Hunan Normal University, College of Physical Education

IPD SHARING:
Plan to Share IPD: No
IPD protocol was not submitted in the approved institutional review board protocol.